CLINICAL TRIAL: NCT03370640
Title: A 2-Part Ascending Multiple Oral Dose, Open-Label Study Assessing the Safety, Tolerability, and Pharmacokinetics of SEP-363856 in Japanese Male and Female Subjects With Schizophrenia.
Brief Title: Study Assessing the Safety, Tolerability, and Pharmacokinetics of SEP-363856 in Japanese Male and Female Subjects With Schizophrenia in 2 Parts (Part 1 and 2).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DA801004; JapicCTI-173787 (Registry Identifier: JAPIC ClinicalTrials Information)
Record Dates: First submitted 2017-11-22; First posted 2017-12-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- SEP-363856 Part 1 Cohort 1 (Experimental): An oral 25 mg dose of SEP 363856 once daily for 3 days, then 50 mg dose of SEP-363856 once daily for 7 days.
  Interventions: Drug: SEP-363856
- SEP-363856 Part 1 Cohort 2 (Experimental): An oral 50 mg dose of SEP 363856 once daily for 3 days, then 75 mg dose of SEP-363856 once daily for 7 days.
  Interventions: Drug: SEP-363856
- SEP-363856 Part 2 Cohort 3 (Experimental): An oral 25 mg dose of SEP 363856 once daily for 3 days, 50 mg dose of SEP 363856 once daily for 4 days, and then 75 mg dose of SEP-363856 once daily for 7 days.
  Interventions: Drug: SEP-363856

INTERVENTIONS:
Drug: SEP-363856 — An oral 25 or 50mg dose of SEP 363856

SUMMARY:
This is a multiple oral dose, open-label study to assess the safety, tolerability, and pharmacokinetics of SEP-363856 in Japanese subjects with schizophrenia.

DETAILED DESCRIPTION:
This multicenter study will be conducted in 2 parts (Part 1 and 2). This is an ascending multiple oral dose, open-label study assessing the safety, tolerability, and pharmacokinetics of SEP-363856 in male and female subjects with schizophrenia. In part 1, subjects will have up to two visits, including a screening visit, and a 17-day in-clinic period. Eligible subjects will be admitted to the clinic on Day -4 to start or complete a taper/washout of their prior antipsychotic medication(s) under the supervision of the Investigator. On Day 1, after subjects have successfully completed the taper/washout of prior medication, subjects will be administered SEP 363856, and dosing with SEP 363856 will continue once-daily for 10 days in-clinic dosing. From Day 11 through Day 13, inclusive, subjects will be restabilized on their adequate antipsychotic medication(s) before clinic discharge on Day 14. Some subjects may require a longer restabilization process based on Investigator judgment. Subjects who discontinue the study prior to Day 13 will require an in-clinic stay for 3 days (or longer based on Investigator judgment) for restabilization on prior medications. In Part 2, Subjects will have up to two visits, including a screening visit, and a 21-day in-clinic period. Eligible subjects will be admitted to the clinic on Day -4 to start or complete a taper/washout of their prior antipsychotic medication(s) under the supervision of the Investigator. On Day 1, after subjects have successfully completed the taper/washout of prior medication, subjects will be administered SEP 363856, and dosing with SEP 363856 will continue once-daily for 14 days in-clinic dosing. From Day 15 through Day 17, inclusive, subjects will be restabilized on their adequate antipsychotic medication(s) before clinic discharge on Day 18. Some subjects may require a longer restabilization process based on Investigator judgment. Subjects who discontinue the study by Day 17 will require an in-clinic stay for 3 days (or longer based on Investigator judgment) for restabilization on prior medications.

ELIGIBILITY:
Inclusion Criteria:The subjects who fulfill the following criteria will be included in the study.

* Subjects who are fully informed of and understand the objectives, procedures, and possible benefits and risks of the study and who voluntarily provide written consent to participate in the study. If the subject is considered a minor or is hospitalized involuntarily at the time of collection of the informed consent, written consent will be obtained from a legally acceptable representative (guardian) in addition to that obtained from the subject.
* Japanese subject with schizophrenia between 18 to 55 years of age at the time of consent.
* Subject who has schizophrenia diagnosed by Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5), diagnostic criteria, and in the opinion of the Investigator has been clinically stable.
* Subject who has body weight ≥ 40.0 kg and body mass index (BMI) ≥ 18.5 (BMI = body weight [kg] / [height (m)]2).
* Female subjects who are premenopausal and of childbearing potential must have a negative serum pregnancy test result at screening, and a negative urine pregnancy test result at clinic admission (Note: Positive urine pregnancy test will be confirmed by serum pregnancy test). Subjects who are not pregnant and are not nursing mothers.
* Female subjects who are of childbearing potential and male subjects whose partners are of childbearing potential must agree to use adequate and appropriate contraception throughout the study starting the day obtaining informed consent and for at least 30 days after the last study drug administration.
* Subjects who are able to comply with the study requirements, including physical examination, assessments, and reporting symptoms.

Exclusion Criteria:The subjects who meet any of the following criteria will be excluded from the study.

* Subject experienced an acute exacerbation of psychiatric symptoms requiring change in antipsychotic medication (with reference to drug or dose) within 3 months before screening.
* Subjects who received any sustained-release formulation (depot preparation) of antipsychotic medications within 3 months before screening.
* Subjects who received electroconvulsive therapy within 3 months before screening or is expected to require ECT during the study.
* Subjects has a history of alcohol or substance related disorders (according to DSM-5 criteria) within 6 months before screening or a positive urine drug screen at screening.
* Subjects who received other investigational products or post-marketing clinical study drugs within 3 months before screening or who have enrolled in but have not completed another clinical or post-marketing study before screening.
* Subjects with a history or complication (s) of malignant tumor within 5 years before screening, except for adequately treated basal cell or squamous cell carcinoma of skin or cervix carcinoma in situ.
* Subjects are considered by the Investigator to be affected by potent central nervous system depressants (including barbiturate).
* Subjects have previous or existing infection with HIV at screening. Subjects have a positive test for Syphilis serum reaction, Hepatitis B surface antigen or Hepatitis C antibody at screening.
* Subjects with specific suicidal ideation or those with a suicide attempt history
* Subjects have any clinically significant unstable medical condition or any clinically significant chronic disease that in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in the study, etc

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs), serious adverse events (SAEs), and AEs resulting in study discontinuation. | Two weeks in part 1, 3 weeks in part 2.
  adverse events (AEs), serious adverse events (SAEs), and AEs resulting in study discontinuation.

SECONDARY OUTCOMES:
Plasma concentrations of SEP-363856 and its metabolite SEP-363854 | Twelve days in part 1, 16 days in part 2.
  Plasma concentration ( Day -1 , Day 1, Day 10, and Day 11) in part 1, plasma concentration ( Day -1 , Day 1, Day 14, and Day 15) in part 2.

CONTACTS AND LOCATIONS:
Locations (8):
- Japan (8):
  - Hotei Hospital, Kōnan, Aichi-ken
  - Soushu Hospital, Atsugi, Kanagawa
  - Mental Support SOYOKAZE Hospital, Ueda, Nagano
  - Asakayama General Hospital, Sakai, Osaka
  - Showa University Karasuyama Hospital, Setagaya-Ku, Tokyo
  - Narimasu Kosei Hospital, Itabashi-Ku
  - Yuge Hospital, Kumamoto
  - National Hospital Organization Hizen Psychiatric Center, Saga